CLINICAL TRIAL: NCT02142062
Title: Prospective, Single-arm, Multi-center, Pilot Study of IVUS Imaging Used as an Adjunct to Multiplanar Venography During Iliac-common Femoral Vein Assessment for Possible Endovascular Intervention
Brief Title: Venogram vs. Intravascular Ultrasound (IVUS) for Diagnosing Iliac Vein Obstruction
Acronym: VIDIO
Status: Completed | Type: Observational
Sponsor: Volcano Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 007-13
Record Dates: First submitted 2014-05-14; First posted 2014-05-20 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Iliac Venous Compression
Keywords: Venous outflow obstruction; Iliac Vein; Common Femoral Vein; Iliac Compression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Venography and IVUS imaging guiding treatment

SUMMARY:
The purpose of this study is to demonstrate that IVUS identifies more instances of significant iliac and common femoral vein outflow obstruction than multiplanar venography.No hypothesis testing is planned.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be > 18 and < 85 years of age
* Willing to participate in and able to understand, read and sign the informed consent document before the planned procedure
* CEAP clinical classification: C4, C5, or C6 (enrollment of C4 and C5 subjects will be capped at 50, such that at least 50 C6 subjects can be enrolled)
* On duplex ultrasound: patent common femoral vein, and patent deep femoral vein, and/or femoral vein of the study leg
* Undergoing iliofemoral and inferior vena caval venography with the intent to treat obstructive lesions

Exclusion Criteria:

* Subject cannot or will not provide written informed consent
* Previous venous stent implantation involving the study leg or inferior vena cava
* Previous venovenous bypass surgery involving the study leg
* Known metal allergy precluding endovascular stent implantation
* Known reaction or sensitivity to iodinated contrast that cannot be managed with premedication
* Subjects who are pregnant (women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment
* Severe, untreated (and readily treatable) superficial venous reflux (great saphenous vein >7 mm in diameter, and/or small saphenous vein >4 mm in diameter)
* Acute deep venous thrombosis involving either leg
* Known history of chronic total occlusion of the common femoral vein of the study leg.
* Known history of thrombophilia (e.g., protein C or S deficiency, anti-thrombin III deficiency, presence of lupus anticoagulant, etc.)
* Venous compression caused by tumor encasement
* Venous outflow obstruction caused by tumor thrombus
* Life expectancy of less than 6 months
* Elevated baseline blood creatinine (value greater than the upper limit of the normal range)
* Any concurrent disease or condition that, in the opinion of the Investigator, would make the subject unsuitable for participation in the study; examples include but are not limited to the inability to lie supine for the index procedure (e.g., severe congestive heart failure), thrombocytopenia or other hematological disorders associated with an unacceptable risk of bleeding, implanted orthopedic hardware that precludes proper imaging, etc.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with iliac compression disease CEAP classification 4-6. Hospitals, venous clinics
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
100 patients with Clinical-Etiologic-Anatomic-Pathophysiologic (CEAP) classification C4-6 undergoing iliac and common femoral and venography with intention to treat venous outflow obstruction. | 6 month
  Primary Endpoints: Both venous IVUS and traditional venography will provide measurements of minimum and maximum diameter reduction due to iliofemoral venous obstruction/compression; cross-sectional area reduction will also be measured by IVUS, and calculated for venography (from min. and max. diameters, assuming elliptical cross-section6). The diameters and cross-sectional area are compared to adjacent reference vessel in order to calculate the degree of stenosis. The percentage of significant stenosis detected at various thresholds [e.g., 50%, 60%, 70%, 80%, for diameter reduction, and (separately) for area reduction] with each method will be compared in a pair-wise fashion. This will be done with descriptive statistics of the detection rates for each method, and the rate of discordance between the two. In addition to the binary outcome of significant stenosis, the numeric values for diameters and cross-sectional areas will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gagne, M.D., Principal Investigator — Southern Connecticut Vascular Center
Locations (14):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - Arizona Heart, Phoenix, Arizona
  - Southern CT Vascular Center, Bridgeport, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Vein Center of Southwest Louisiana/Imperial Health, Lake Charles, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - The Mount Sinai Medical Center, New York, New York
  - SUNY Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Allegheny Vein and Vascular Clinic, Bradford, Pennsylvania
- Hesperia Hospital, Modena, Italy
- Szpital Kliniczny Przemienienia Pańskiego, Poznan, Poznan, Poland
- St Thomas Hospital, London, United Kingdom

REFERENCES:
- [Background] Murad MH, Coto-Yglesias F, Zumaeta-Garcia M, Elamin MB, Duggirala MK, Erwin PJ, Montori VM, Gloviczki P. A systematic review and meta-analysis of the treatments of varicose veins. J Vasc Surg. 2011 May;53(5 Suppl):49S-65S. doi: 10.1016/j.jvs.2011.02.031. PMID 21536173
- [Background] Bergan JJ, Schmid-Schonbein GW, Coleridge Smith PD, Nicolaides AN, Boisseau MR, Eklof B. Chronic venous disease. Minerva Cardioangiol. 2007 Aug;55(4):459-76. No abstract available. English, Italian. PMID 17653022
- [Background] Raju S, Neglen P. Clinical practice. Chronic venous insufficiency and varicose veins. N Engl J Med. 2009 May 28;360(22):2319-27. doi: 10.1056/NEJMcp0802444. No abstract available. PMID 19474429
- [Background] Neglen P, Raju S. Intravascular ultrasound scan evaluation of the obstructed vein. J Vasc Surg. 2002 Apr;35(4):694-700. doi: 10.1067/mva.2002.121127. PMID 11932665
- [Background] Raju S, Neglen P. High prevalence of nonthrombotic iliac vein lesions in chronic venous disease: a permissive role in pathogenicity. J Vasc Surg. 2006 Jul;44(1):136-43; discussion 144. doi: 10.1016/j.jvs.2006.02.065. PMID 16828437
- [Background] Murphy EH, Broker HS, Johnson EJ, Modrall JG, Valentine RJ, Arko FR 3rd. Device and imaging-specific volumetric analysis of clot lysis after percutaneous mechanical thrombectomy for iliofemoral DVT. J Endovasc Ther. 2010 Jun;17(3):423-33. doi: 10.1583/10-3088.1. PMID 20557187
- [Background] Raju S. Best management options for chronic iliac vein stenosis and occlusion. J Vasc Surg. 2013 Apr;57(4):1163-9. doi: 10.1016/j.jvs.2012.11.084. Epub 2013 Feb 20. PMID 23433816
- [Background] Alhalbouni S, Hingorani A, Shiferson A, Gopal K, Jung D, Novak D, Marks N, Ascher E. Iliac-femoral venous stenting for lower extremity venous stasis symptoms. Ann Vasc Surg. 2012 Feb;26(2):185-9. doi: 10.1016/j.avsg.2011.05.033. Epub 2011 Oct 22. PMID 22018502
- [Background] Vasquez MA, Rabe E, McLafferty RB, Shortell CK, Marston WA, Gillespie D, Meissner MH, Rutherford RB; American Venous Forum Ad Hoc Outcomes Working Group. Revision of the venous clinical severity score: venous outcomes consensus statement: special communication of the American Venous Forum Ad Hoc Outcomes Working Group. J Vasc Surg. 2010 Nov;52(5):1387-96. doi: 10.1016/j.jvs.2010.06.161. Epub 2010 Sep 27. PMID 20875713
- [Background] Stacey MC, Burnand KG, Layer GT, Pattison M, Browse NL. Measurement of the healing of venous ulcers. Aust N Z J Surg. 1991 Nov;61(11):844-8. doi: 10.1111/j.1445-2197.1991.tb00169.x. PMID 1750819
- [Background] Eklof B, Rutherford RB, Bergan JJ, Carpentier PH, Gloviczki P, Kistner RL, Meissner MH, Moneta GL, Myers K, Padberg FT, Perrin M, Ruckley CV, Smith PC, Wakefield TW; American Venous Forum International Ad Hoc Committee for Revision of the CEAP Classification. Revision of the CEAP classification for chronic venous disorders: consensus statement. J Vasc Surg. 2004 Dec;40(6):1248-52. doi: 10.1016/j.jvs.2004.09.027. PMID 15622385
- [Derived] Gagne PJ, Gasparis A, Black S, Thorpe P, Passman M, Vedantham S, Marston W, Iafrati M. Analysis of threshold stenosis by multiplanar venogram and intravascular ultrasound examination for predicting clinical improvement after iliofemoral vein stenting in the VIDIO trial. J Vasc Surg Venous Lymphat Disord. 2018 Jan;6(1):48-56.e1. doi: 10.1016/j.jvsv.2017.07.009. Epub 2017 Oct 13. PMID 29033314
- [Derived] Gagne PJ, Tahara RW, Fastabend CP, Dzieciuchowicz L, Marston W, Vedantham S, Ting W, Iafrati MD. Venography versus intravascular ultrasound for diagnosing and treating iliofemoral vein obstruction. J Vasc Surg Venous Lymphat Disord. 2017 Sep;5(5):678-687. doi: 10.1016/j.jvsv.2017.04.007. Epub 2017 Jun 28. PMID 28818221